CLINICAL TRIAL: NCT01364376
Title: S-1 Plus Oxaliplatin Compared With Fluorouracil, Leucovorin Calcium Plus Oxaliplatin as Perioperative Chemotherapy for Advanced Gastric Carcinoma: a Multi-center, Open-labeled, Randomized Controlled Trial
Brief Title: S-1 Plus Oxaliplatin Compared With Fluorouracil, Leucovorin Calcium Plus Oxaliplatin as Perioperative Chemotherapy for Advanced Gastric Carcinoma
Acronym: Focus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Jiren Yu, Chief doctor, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZYYY-GC1105
Record Dates: First submitted 2011-05-19; First posted 2011-06-02 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Stomach Neoplasms
Keywords: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — S 1 (combination); Oxaliplatin; Fluorouracil; Leucovorin

ARMS (2):
- FOLFOX (Active Comparator)
  Interventions: Drug: S-1; Oxaliplatin; 5-Fu; Leucovorin Calcium
- SOX (Experimental)
  Interventions: Drug: S-1; Oxaliplatin; 5-Fu; Leucovorin Calcium

INTERVENTIONS:
Drug: S-1; Oxaliplatin; 5-Fu; Leucovorin Calcium — FOLFOX:
  oxaliplatin 130mg/m2 on day 1, CF 400mg/m2 on day 1, 5-Fu 400mg/m2 on day 1; 5-FU 2400 mg/m2 46hr civ regimen repeated every 3 weeks Pre-operative chemotherapy: 2-4 cycles and peri-operative chemotherapy consist of 6 cycles
  SOX:
  oxaliplatin 130mg/m2 on day 1, S-1 for 14 days regimen repeated every 3 weeks Pre-chemotherapy: 2-4 cycles, totally 6 cycles of perioperative chemotherapy

SUMMARY:
This is a randomized multicenter controlled study of oxaliplatin, leucovorin calcium , plus 5-fluorouracil (FOLFOX) compared with S-1 plus oxaliplatin (SOX) as perioperative chemotherapy for advanced gastric cancer.

Hypothesis: SOX is not inferior to FOLFOX as perioperative chemotherapy for advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed gastric adenocarcinoma,diagnosed as locally advanced gastric cancer and primary tumor invades or penetrates serosa
* Ambulatory males or females, aged 18-80 years old
* ECOG score 0-2
* Given informed consent
* Life expectancy more than 3 months
* Measurable lesion
* Normal cardiac, hepatic, renal, and bone marrow function(WBC:3.5×10^9/l~12×10^9/l;PLT:>100×109/l;Bil:<1.5 fold of upper limit value; ALT/AST:<2.5 fold of upper limit value;Ccr:>80ml/min;Cr:1.5mg/dl)

Exclusion Criteria:

* Prior stomach surgery
* Previous cytotoxic chemotherapy, radiotherapy, target therapy or immunotherapy for any tumor
* History of another malignancy except cured basal cell carcinoma of skin and cured carcinoma in-situ of uterine cervix
* distant metastasis(such as No.16 and No.13 lymphnode,liver, lung,brain,bones or peritoneal metastasis)
* Severe bleeding
* Bowel obstruction, ileus or complete pyloric obstruction
* Serious uncontrolled concomitant disease
* History of myocardial infarction in 6 months
* Woman with on-going pregnancy or breast-feeding, or contemplating pregnancy
* Systemic treatment with corticosteroid
* Patients judged inappropriate for the trial by the physicians

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 583 (Actual)
Dates: Start 2011-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
overall survival | 3-year

SECONDARY OUTCOMES:
progression-free survival(PFS) | 3-year
clinical response | 6 or 12 weeks
pathological response | within 10 days after surgery
Number of Participants with grade 3/4 adverse Events | 6 Years

CONTACTS AND LOCATIONS:
Overall Officials: Jiren Yu, Principal Investigator — The First Affiliated Hospital of Medical School of Zhejiang University
Locations (8):
- China (8):
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Medical School of Zhejiang University, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Medical School of Zhejiang University, Hangzhou, Zhejiang
  - Jiaxing First Hospital, Jiaxing, Zhejiang
  - Ningbo Medical Treatment Center Lihuili Hospital, Ningbo, Zhejiang
  - The second affiliated hospital of Wenzhou medical college, Wenzhou, Zhejiang

REFERENCES:
- [Derived] Yu J, Gao Y, Chen L, Wu D, Shen Q, Zhao Z, Liu W, Yang H, Zhang Q, Wang X, Hu P, Zheng Z, Wang X, Liu H, Xu Z, Yan Z, Wu Y, Jin M, Zhang Q, Liu X, Zhu K, Shou C. Effect of S-1 Plus Oxaliplatin Compared With Fluorouracil, Leucovorin Plus Oxaliplatin as Perioperative Chemotherapy for Locally Advanced, Resectable Gastric Cancer: A Randomized Clinical Trial. JAMA Netw Open. 2022 Feb 1;5(2):e220426. doi: 10.1001/jamanetworkopen.2022.0426. PMID 35226081